CLINICAL TRIAL: NCT05663021
Title: Feasibility in Identification of Suitable Candidates for Elimination of Axillary Surgery in Breast Cancer Patients With Initial Biopsy-confirmed Nodal Metastases
Brief Title: Feasibility in Identification of Breast Cancer Candidates for Elimination of Axillary Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Director of Department of Breast Surgery, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FIERCE
Record Dates: First submitted 2022-12-14; First posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Breast Cancer
Keywords: neoadjuvant chemotherapy; nodal response; core needle biopsy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrasound-Guided Biopsy of Tumor Site during neoadjuvant chemotherapy (Experimental): For patients who were not evaluated as progressive disease by the latest imaging measurement, repeated CNB (RCNB) was performed after 2-4 cycles of NAC, depending on the total cycles of NAC. Tissue is acquired from different sections of the lesion from different angles to minimize the impact of tumor heterogeneity. For each patient, 3 to 4 tissue specimens are collected and sent for pathological review to examine whether there is residual malignancy (residual cancer, pleomorphic tissue) in the tumor site that is tattooed.
  Interventions: Diagnostic Test: Ultrasound-guided core needle biopsy in breast

INTERVENTIONS:
Diagnostic Test: Ultrasound-guided core needle biopsy in breast — For patients who were not evaluated as progressive disease by the latest imaging measurement, repeated core needle biopsy is conducted within the baseline tattooed area after 2 to 4 cycles of neoadjuvant chemotherapy, depending on the total cycles of chemotherapy. Tissue is acquired from different sections of the lesion from different angles to minimize the impact of tumor heterogeneity. For each patient, 3 to 4 tissue specimens are collected and sent for pathological review to examine whether there is residual malignancy (residual cancer, pleomorphic tissue) in the tumor site that is tattooed.

SUMMARY:
Preoperative identification of patients with pathologic complete response or residual disease in axilla can aid in tailoring subsequent axillary surgery including omission of axillary surgery based on tumor biology and response to neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVE:

To determine the accuracy of on-treatment core needle biopsy in breast to predict nodal response after neoadjuvant chemotherapy.

OUTLINE:

Early breast cancer patients aged above 18 and below 70 years with biopsy-confirmed, clinically T1-4, N1-3, and M0 disease are eligible for this study. Breast cancer is proven pathologically in all patients using the baseline core needle biopsy, and the skin of all patients is tattooed at the baseline. Metastatic lymph nodes are diagnosed with core needle biopsy or fine needle aspiration. All the patients undergo clip placement into node with biopsy-confirmed metastases at the time of diagnosis. For patients who were not evaluated as progressive disease by the latest imaging measurement, repeated CNB (RCNB) was performed after 2-4 cycles of NAC, depending on the total cycles of NAC., repeated core needle biopsy is conducted within the baseline tattooed area after 2 to 4 cycles of neoadjuvant chemotherapy, depending on the total cycles of chemotherapy. Tissue is acquired from different sections of the lesion from different angles to minimize the impact of tumor heterogeneity. For each patient, 3 to 4 tissue specimens are collected and sent for pathological review to examine whether there is residual malignancy (residual cancer, pleomorphic tissue) in the tumor site that is tattooed.

All the patients receive planned axillary surgery after completion of neoadjuvant chemotherapy. the surgical approach was determined by the treating breast surgical oncologist including targeted axillary dissection (TAD) or axillary lymph node dissection, mainly based on the intraoperative TAD results

PROJECTED ACCRUAL: A total of 180 patients will be accrued for this study within 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical stage T1-4 N1-3M0 breast cancer at diagnosis (prior to neoadjuvant chemotherapy) by American Joint Committee on Cancer (AJCC) staging 7th edition
2. Aged above 18 and below 70 years
3. No other malignancy within 5 years of registration with the exception of basal cell or squamous cell carcinoma of the skin treated with local resection only or carcinoma in situ of the cervix
4. Patients must have had estrogen receptor, progesterone receptor and HER2 status (by immunohistochemistry [IHC] and/or in situ hybridization [ISH]) evaluated on core needle biopsy prior to starting neoadjuvant chemotherapy
5. Completing all planned cycles and regimens of neoadjuvant chemotherapy followed by axillary surgery

Exclusion Criteria:

1. Nonrepresentative core needle biopsy in the breast during neoadjuvant chemotherapy
2. Inflammatory breast cancer

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female breast cancer patients are enrolled
Enrollment: 191 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2021-06-26 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Diagnostic Accuracy of Ultrasound-Guided Core Biopsy of Initial Breast Cancer Region Compared to Axillary Surgery with Pathologic Evaluation Cancer Region Compared to Standard Surgery with Pathologic Evaluation | 1 day
  Accuracy of core biopsy determined by biopsy results to the axillary pathologic evaluation removed during standard surgery. Estimates and 95% confidence intervals for accuracy, sensitivity, false negative rate (FNR), specificity as well as the negative predictive value (NPV) reported for FNA and core biopsy based on the exact Clopper-Pearson method.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhi-Min Shao, Shanghai, Shanghai Municipality, China